CLINICAL TRIAL: NCT03777904
Title: The Iron Content of Ferritin in Serum and Urine of Children With High Serum Ferritin Levels
Status: Terminated | Type: Observational
Why Stopped: Analysis of first 11 subjects resulted in values that were too varied to make the study feasible.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 00117617
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Iron Overload
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with high serum ferritin: Children with very high serum ferritin levels and confirmed iron toxicity will have a urine sample and blood sample drawn at the same time. Both samples will have ferritin levels and iron content measured and compared for correlation.
  Interventions: Diagnostic Test: Serum Ferritin level; Diagnostic Test: Serum Ferritin iron content; Diagnostic Test: Urine Ferritin level; Diagnostic Test: Urine ferritin iron content

INTERVENTIONS:
Diagnostic Test: Serum Ferritin level — Serum ferritin level will be collected with other clinical labs and measured in the research lab
Diagnostic Test: Serum Ferritin iron content — Blood will be collected with other clinical labs and the iron content in the ferritin will be measured in the research lab
Diagnostic Test: Urine Ferritin level — Urine will be collected non-invasively and analyzed for ferritin level
Diagnostic Test: Urine ferritin iron content — Urine will be collected non-invasively and analyzed for iron content within the ferritin

SUMMARY:
A serum ferritin level can reflect the total body iron content, thus a very low serum ferritin is commonly used as an indicator of iron deficiency and a very high serum ferritin is commonly used as a marker of iron overload. Ferritin is a shell of protein in which iron is stored. Ferritin is an acute phase reactant, and serum ferritin levels can increase during inflammatory conditions. Consequently, an elevated ferritin level might mean there is an excess of storage iron, or might simply mean that inflammation has resulted in high levels of the ferritin shell, containing little iron.

The research team is able to quantify the amount of iron in ferritin using inductively conducted plasma mass spectrometry, in the Heme and Iron Core Laboratory at the University of Utah. Thus, it can be determined whether in a child with a very high serum ferritin level, that ferritin is loaded with iron or is actually very low in iron. Neonates and young children with certain liver disorders characteristically have a very high serum ferritin level. These conditions are gestational alloimmune liver disease (GALD) and hemophagocytic lymphohistiocytosis (HLH). It is not clear what the iron content of the ferritin is in these neonates. Knowing this will be a step toward understanding whether the pathogenesis of these conditions involves iron overload. Additionally, if urine ferritin and iron levels correlate with serum ferritin and iron levels, urine may be used as a non-invasive way to monitor iron status.

In this study, serum and urine samples will be collected from children with high serum ferritin levels and confirmed iron toxicity. Both ferritin and iron content within ferritin will be measured in the serum and urine samples and compared for correlation.

ELIGIBILITY:
Inclusion Criteria:

* Children with ferritin levels > 1000 ng/mL

Exclusion Criteria:

* None

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with high ferritin levels and confirmed iron toxicity.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Correlation of serum and urine ferritin levels | 1 year
  Serum levels of ferritin will be compared to urine ferritin levels to evaluate whether urine can be used to calculate ferritin levels in the body non-invasively
Correlation of iron content within serum and urine ferritin levels | 1 year
  Serum iron content of ferritin will be compared to urine iron content of ferritin levels to evaluate whether urine can be used to calculate total body iron content non-invasively

CONTACTS AND LOCATIONS:
Overall Officials: Robert Christensen, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Hospital, Salt Lake City, Utah, United States